CLINICAL TRIAL: NCT07067242
Title: Prevalence of Cervicogenic Headache Among Lab Technicians
Brief Title: Prevalence of Cervicogenic Headache in Lab Technicians
Status: Completed | Type: Observational
Sponsor: Elite College of Management Sciences, Gujranwala, Pakistan (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-GCUF079345
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic headache; Posture; Neck pain; Lab technicians
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to determine the prevalence of cervicogenic headache among lab technicians

DETAILED DESCRIPTION:
Cervicogenic headache is a type of headache characterized by chronic hemi- cranial pain referred to the head from either the cervical spine or soft tissues within the neck .It reduces the quality of life .

Objective: The objective of this study is to determine the prevalence of cervico-genic headache among lab technicians in Gujranwala.

ELIGIBILITY:
Inclusion Criteria:

Sitting duration of 3 or more than 3 hours Having neck pain for atleast1 month Consistant Unilateral headache Age 30 to 44

Exclusion Criteria:

Recent fracture Recent surgery Congenital conditions of cervical spine History of traumatic neck injuries or cervical spine surgery. Diagnosis of primary headache disorders (e.g., migraines, tension-type headaches).(21)

Ages: 30 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Lab technicians of Gujranwala
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4th week
  To measure pain
Self prepared questionnaire | 4th week
  To measure Cervicogenic headache associated disability

CONTACTS AND LOCATIONS:
Overall Officials: Rukhma Mauzzam, Principal Investigator — Elite College of Management Science
Locations (1):
- Private and public labs of Gujranwala, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young IA, Dunning J, Butts R, Cleland JA, Fernandez-de-Las-Penas C. Psychometric properties of the Numeric Pain Rating Scale and Neck Disability Index in patients with cervicogenic headache. Cephalalgia. 2019 Jan;39(1):44-51. doi: 10.1177/0333102418772584. Epub 2018 Apr 19. PMID 29673262
- [Background] Sjaastad O, Bakketeig LS. Prevalence of cervicogenic headache: Vaga study of headache epidemiology. Acta Neurol Scand. 2008 Mar;117(3):173-80. doi: 10.1111/j.1600-0404.2007.00962.x. Epub 2007 Nov 20. PMID 18031563
- [Background] Knackstedt H, Bansevicius D, Aaseth K, Grande RB, Lundqvist C, Russell MB. Cervicogenic headache in the general population: the Akershus study of chronic headache. Cephalalgia. 2010 Dec;30(12):1468-76. doi: 10.1177/0333102410368442. Epub 2010 May 19. PMID 20974607
- [Background] 18. Kanniappan, V., Abraham, S. S., & Veeragoudhaman, T. S. (2022). PREVALENCE OF CERVICOGENIC HEADACHE AMONG YOUNG POPULATION. International Journal of Research-GRANTHAALAYAH, 10(9), 14-26.
- [Background] Almesned IS, Alqahtani NG, Alarifi JA, Alsaawy TN, Agha S, Alhumaid MA. Prevalence of primary headache among medical students at King Saud bin Abdulaziz University for Health Sciences, Riyadh, Saudi Arabia. J Family Med Prim Care. 2018 Nov-Dec;7(6):1193-1196. doi: 10.4103/jfmpc.jfmpc_240_18. PMID 30613496
- [Background] Muayqil T, Al-Jafen BN, Al-Saaran Z, Al-Shammari M, Alkthiry A, Muhammad WS, Murshid R, Alanazy MH. Migraine and Headache Prevalence and Associated Comorbidities in a Large Saudi Sample. Eur Neurol. 2018;79(3-4):126-134. doi: 10.1159/000487317. Epub 2018 Mar 14. PMID 29539610
- [Background] 10. Mathur, R., & Tegh, S. S. A Cross-Sectional Study on the Prevalence of Cervicogenic Headache Amongst University Students.
- [Background] Fortner MO, Woodham TJ, Oakley PA, Harrison DE. Is the cervical lordosis a key biomechanical biomarker in cervicogenic headache?: a Chiropractic Biophysics(R) case report with follow-up. J Phys Ther Sci. 2022 Feb;34(2):167-171. doi: 10.1589/jpts.34.167. Epub 2022 Feb 23. PMID 35221522
- [Background] Racicki S, Gerwin S, Diclaudio S, Reinmann S, Donaldson M. Conservative physical therapy management for the treatment of cervicogenic headache: a systematic review. J Man Manip Ther. 2013 May;21(2):113-24. doi: 10.1179/2042618612Y.0000000025. PMID 24421621
- [Background] Al Khalili Y, Ly NK, Murphy PB. Cervicogenic Headache. 2022 Oct 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507862/ PMID 29939639
- [Background] Barmherzig R, Kingston W. Occipital Neuralgia and Cervicogenic Headache: Diagnosis and Management. Curr Neurol Neurosci Rep. 2019 Mar 19;19(5):20. doi: 10.1007/s11910-019-0937-8. PMID 30888540